# TRANSCENDENCE RESEARCH: Holistic Education For Colonized Countries Primarily English Speaking

NCT06098755

January 24, 2026

#### **Brief Summary**

This Intervention study (also called experimental study) emphasizes active listening skills to understand participant preferences. The purpose is to provide cost-effective pastoral counseling for stress management in both workplace and everyday life. The eligibility requirement has been updated to include UNMARRIED Couples, Bachelor, and Bachelorette Alaska Medicaid recipients age 22 and older. The HUMANITARIAN VETERANS ASSOCIATION serves as the tax-exempt peer-review board and liaison for this study.

#### **Detailed Description**

The Headmistress or Headmaster functions as a licensed referral, ordering, and Holistic Medicine prescribing provider only. While tools such as massage chairs may provide immediate stress relief, this study emphasizes economical and sustainable methods of emotional adjustment and self-help practices. The holistic approach focuses on the "Whole Person" concept, incorporating biofeedback to support wellness, healing, and recovery. Biofeedback (i.e. Pulse MD finger monitor, Portable automatic blood pressure wrist monitor, Contactless infrared thermometer) tools are used to document the most recent vital signs. Facility parking availability and rules must be explained in print before the appointment.

## Scheduled Initial Overnight Natural Observation, Here and Now Psychotherapy and Initial Assessment

An initial overnight Natural Observation is required to validate study accuracy. New patients are expected to demonstrate self-control exceeding the standards of the Irresistible Impulse Test. Specific indicators for recidivism and serious mental health concerns—such as signs of deviant behavior, lack of self-control, poor hygiene, or inappropriate sexual conduct—must be documented. During the scheduled overnight Natural Observation, Virtual Tribunal Monastery utilizes "Here and Now" psychotherapy focusing on present feelings and interpersonal reactions during sessions. For these treatments, most recent vital signs are documented.

#### **Appointment Itinerary**

- 1. Identification and Consent Show identification in person. Review and confirm mutual terms of agreement in print on consent forms
- 2. Tour of Nonclinical Setting portable toilet for each patient ( 5 U.S. gallon bucket wi/lid, portable toilet seat, bottled water, wipes, sanitizer, and scented trash bags).
- 3. Opening Prayer Philippians 4:4-9 (KJV)

- 4. Document vital signs
- 5. Bible Study listen to the full audiobook WITNESS TO HOPE, THE BIOGRAPHY OF POPE JOHN PAUL II, GEORGE WEIGEL

#### **Church and Appointment Policies**

Please remind all patients that the Church maintains a strict no-smoking policy on the premises. If a patient leaves before an appointment is concluded, the session is terminated. The patient must then either reschedule for a full new appointment or be referred to services best suitable to their needs or preferences.

#### Safety and Security

Ensure all indoor floodlights are set to motion detection. Furthermore, a police report must be filed with tangible evidence for every incident as it occurs. This includes reporting any suspected human trafficking, stalking, or harassment involving unknown or violent female repeat offenders.

#### **During the Scheduled Initial Overnight Natural Observation**

A controlled area, Security & Access: often defined as areas under surveillance, requiring authorized access or escorts, such as in government or high-security facilities, involves the usage of a portable toilet including not leaving the controlled area until the appointment is complete. One portable toilet for each person includes a bucket w/lid, toilet seat and disposable scented trash bags to dispose of waste off premises. Patients are encouraged to bring an overnight bag with wet wipes, alcohol, vaseline, a towel, pillow, clean clothes, pajamas, t-shirt, underwear, socks, a few sack lunches, a few bottled waters, and snacks. I also recommend patients bring earplugs for deep meditation practices. The scheduled initial overnight Natural Observation is also intended to provide a safe place for patients to adapt to inevitable norms while practicing maintaining focus without distractions for desensitization techniques: Listening to the complete audiobook WITNESS TO HOPE, THE BIOGRAPHY OF POPE JOHN PAUL II. GEORGE WEIGEL at the public library HOOPLA App on TV. In hostile environments, the patient may notice or become socially-aware of the urge to run away. The appointment may be cancelled at any time for rescheduling or referral to services more suitable to individual needs or preferences. Virtual Tribunal Monastery follows strict safety protocols in Marginalized communities. If watching adult movies, seeing sexually-explicit artwork, Catholicism and seeing a firearm is extremely uncomfortable; the patient will be given options If the patient has additional concerns.

#### Intake Interview Before Providing a Holistic Medicine Prescription...

Psychological and neurological tests are designed to assist with desensitization techniques while helping participants adapt to social norms with inclusive language. The goal is to strengthen objectivity, focus, and resilience against distractions. These assessments support the overall mission of guiding participants toward balance, adaptation, and holistic well-being. A comprehensive case study and treatment plan must be completed. This includes an initial intake interview summarizing the initial overnight Natural Observation to assess the individual or social unit progress. Nonclinical variables, including social determinants and socioeconomic factors, must be classified under Holistic Medicine using the ICD-10 Z-codes (SDOH) Social Determinants of Health.

#### **Conditions of Focus of Study Relevant to Stress Management**

This study emphasizes holistic approaches to stress management by focusing on conditions that commonly affect workplace and daily life balance.

#### Areas of focus

Include: Stress, Job, etc... By addressing these conditions, the study aims to help participants achieve relaxation, strengthen resilience, and develop sustainable coping mechanisms.

#### **Intervention Study Design**

Experimental

#### **Outcome Measures**

To further elaborate about Outcome Measures for Holistic Medicine, nonclinical variables are prioritized by its impact while using the qualitative (in layman's terms quality) method that requires a licensed counselor, pastoral counselor or Holistic Medicine provider to best comprehend and have active listening skills to listen for a self-determination or hypothesis towards resolution of this study for individual clients. For clarification about Holistic Medicine Outcome Measures utilize the Maslow's Hierarchy of Needs Motivation Model as a reference and ask the client questions based on the Hierarchy of Needs to determine, which stage on the Hierarchy of Needs best describes the client and whether or not the client has reached optimum wellness in accordance to the Hierarchy or if the client needs more nonclinical variables to reach optimum wellness. The Qualitative evaluation method, usually associated with SOAP (Subjective, Objective, Assessment, Plan) notes summarizes evidence from instructed methods of data collection, naturalistic observation, and existing records. In contrast to qualitative, quantitative is expressed numerically from formal methods of data collection, systemic, and controlled observation; usually associated with goal-based evaluation or STAR (Situation, Task, Action, Result).

#### **Primary Outcome Measures**

Qualitative evaluation method: summarizes evidence from instructed methods of data collection, naturalistic observation, and existing records; usually associated with SOAP (Subjective, Objective, Assessment, Plan) notes.

#### **Secondary Outcome Measures**

Quantitative evaluation method: is expressed numerically from formal methods of data collection, systemic, and controlled observation; usually associated with STAR (Situation, Task, Action, Result) notes.

#### Importance of Informed Consent Form (ICF) and Release of Information (ROI)

The Informed Consent Form (ICF) ensures patients understand the study's purpose, risks, and benefits before agreeing to participate. The Release of Information (ROI) form authorizes the sharing of patient data with designated individuals or organizations, maintaining confidentiality and compliance with ethical standards. For sensitive testing such as STI and Drug Panel testing, appropriate Sexual Consent Forms are necessary when sexual health information is collected or shared for referral, educational, or informational purposes.

#### **Adult Education Component**

This study includes an Adult Time component for desensitization techniques until the repeated appointment consisting of watching Adult movies causes a non-reaction (no masturbation) while gaining beneficial health-related relief from watching adult content. To complete the sexual consent forms accurately, review the sexual consent form instructions. Please remember, the patient is the Proposer (the person wanting to engage in sexual activity). To confirm, the Proposer will input personal preferences on the sexual consent form. This involves structured sessions where patients may consent to be watched while watching adult-rated movies for naturalistic observation. A completely signed sexual consent form is mandatory for safe sex practices, to encourage healthy lifestyle choices and relationships. To further enhance the sexual education experience, engage in guided discussions about graphic sexual content with input onto the ADULT SEXUAL CRITIQUE FORM: A STRATEGY GUIDE, DETAILED RATING AND FEEDBACK.

#### **Purpose**

- To promote open dialogue about sexual health, relationships, and consent.
- To provide a safe, educational environment for discussing sensitive topics.
- Encourage healthy lifestyle choices and relationships.

This component emphasizes the importance of sexual consent, informed decision-making, and respectful dialogue, aligning with the study's broader goals of stress management, holistic education, and ethical practice.

#### **Consent Requirements**

• **Explicit Consent:** Participants must sign specific consent forms before engaging in Adult activities.

## ADULT SEXUAL CRITIQUE FORM: A STRATEGY GUIDE Detailed Rating and Feedback

#### Introduction

**-:**-1-1

Welcome to the Adult Sexual Critique Form strategy guide! This document will provide insights on how to effectively use the critique form to enhance experiences and provide meaningful feedback. This guide focuses on constructively evaluating adult time, movies, and related aspects. The goal is to promote open communication and improve understanding between partners. Remember, *honesty and respect* are key.

## **Understanding the Form**

The Adult Sexual Critique Form is designed to capture detailed feedback across several key areas. It uses a numbered rating system (1-100) for quantitative assessment and includes sections for qualitative elaboration. Here's a breakdown of each section:

| Field | Description |
|---|---|
| Adult Time | Overall quality of the intimate experience. |
| Movie | If applicable, the adult movie watched. |
| Title | The title of the adult movie, if applicable. |
| Viewing Location | Where the viewing or activity took place. |
| Satisfaction | Your overall contentment with the experience. |
| Peace Disturbances | Any interruptions or distractions encountered. |
| Elaboration (Peace<br>Disturbances) | Detailed description of the peace disturbances. |

Dagawinstian

### **Detailed Section Breakdown**

Let's dive deeper into each section of the form to ensure you're providing comprehensive feedback:

#### 1. Adult Time (Rating 1-100):

This section is for rating the overall quality of the adult time. Consider factors like connection, intimacy, and enjoyment. A higher rating indicates a more positive experience. Use the full range of the scale to accurately reflect your feelings.

#### 2. Movie:

State the adult movie viewed (if any). If no movie was watched, enter 'N/A'.

#### 3. Title:

Enter the title of the movie. If no movie was watched, enter 'N/A'.

#### 4. Viewing Location:

Specify where the activity or viewing took place (e.g., 'Bedroom,' 'Living Room').

#### 5. Satisfaction (Rating 1-100):

Rate your overall satisfaction with the experience. Similar to 'Adult Time,' use the full scale to convey your satisfaction level. This rating should reflect your holistic experience.

#### 6. Peace Disturbances:

Note any interruptions or distractions encountered during the experience (e.g., 'Phone ringing,' 'Loud neighbors'). If there were none, enter 'None'.

#### 7. Elaboration (Peace Disturbances):

If you noted any peace disturbances, use this section to provide a detailed description. Include specifics such as the nature of the disturbance, its duration, and its impact on the experience. For example: 'The phone rang multiple times during the movie, which broke the mood and made it difficult to concentrate.'

#### Sections 8-100: Additional Feedback:

These sections are numbered for potential future expansions or specific focused feedback prompts, or even general comments about other aspects of the encounter. When completing these sections, be as specific and constructive as possible.

## **Tips for Providing Effective Feedback**

- **Be Specific:** Avoid vague statements. Provide concrete examples to illustrate your points.
- **Be Honest:** Authentic feedback is crucial for improvement. Express your true feelings and observations.
- **Be Respectful:** Frame your feedback in a constructive and considerate manner. Focus on improving future experiences.
- **Focus on the Positive:** While constructive criticism is valuable, also highlight aspects you enjoyed. This balanced approach promotes a positive atmosphere.
- **Communicate Openly:** Use the form as a starting point for broader discussions. Encourage dialogue to explore each other's perspectives.

## **Example Completion**

Here's an example of how the form might be completed:

Adult Time: 85Movie: Yes

Title: 'Late Night Fantasies'Viewing Location: Bedroom

• Satisfaction: 90

• Peace Disturbances: None

• Elaboration (Peace Disturbances): N/A

## **Summary**

This strategy guide provides a comprehensive overview of the Adult Sexual Critique Form, detailing each section and offering tips for providing effective feedback. By following these guidelines, you can promote open communication, enhance understanding, and improve future experiences. Remember to approach this process with honesty, respect, and a focus on continuous improvement.